CLINICAL TRIAL: NCT05348902
Title: Locked-in Syndrome Caused by Pulmonary Arteriovenous Malformation: A Case Report
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0138
Record Dates: First submitted 2022-04-10; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2021-10

CONDITIONS: Locked-In Syndrome；Pulmonary Arteriovenous Malformation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: In this study, only cases were collected and reported without any intervention or adverse reactions — In this study, only cases were collected and reported without any intervention or adverse reactions

SUMMARY:
In this case, we report a case of atresia syndrome (LIS), a serious neurological disease caused by pulmonary arteriovenous fistula (PAVM). We present a previously healthy middle-aged woman who developed atresia syndrome after severe pontine infarction due to basilar artery occlusion due to undiagnosed arteriovenous malformation. This report reviewed the medical history, post-admission examination and related literature, and concluded that PAVM should be considered as the cause of implicit stroke, especially in young patients with right-to-left shunt, and should be actively treated.

ELIGIBILITY:
Inclusion Criteria:

* A case of Locked-in syndrome due to pulmonary arteriovenous malformation

Exclusion Criteria:

* Patients or family members objected to the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A patient with locked-in syndrome
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-06-02 (Estimated); Study Completion 2022-06-02 (Estimated)

PRIMARY OUTCOMES:
Locked-in syndrome caused by pulmonary arteriovenous malformation . Check list report | 1month
  A recommendation is made for the treatment and prognosis of patients with severe atresia caused by arteriovenous fistula.

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No